CLINICAL TRIAL: NCT04775316
Title: C2654 - Prospective, International, Multicenter, Observational Study to Evaluate the Clinical Performance and Safety of a Silicone-coated Transparent Postoperative Dressing
Brief Title: Prospective, International, Multicenter, Observational Study to Evaluate the Clinical Performance and Safety of a Silicone-coated Transparent Postoperative Dressing
Status: Terminated | Type: Observational
Why Stopped: site stopped recruiting due to limited personell resources
Sponsor: BSN Medical GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: C2654
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Wounds and Injuries; Skin Diseases
MeSH Terms: conditions — Wounds and Injuries; Skin Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with fragile skin: Patient aged 65 years and older presenting with fragile skin and require wound care of an acute wound (laceration or surgical wound). Siliconized sterile wound dressing will be applied for a treatment period of 7 days.
  Interventions: Device: Leukomed T / Tplus skin sensitive treatment

INTERVENTIONS:
Device: Leukomed T / Tplus skin sensitive treatment — Application of sterile wound dressing.

SUMMARY:
Although, a huge number of acute wounds is treated successfully every year, Health Care Professionals (HCPs) are facing more and more problems when treating skin damages or surgical incisions: The number of patients with fragile and/or sensitive skin is highly increasing. Such patients are having a skin integrity issue, meaning the skin is vulnerable to injury, often damaged, or unable to heal.

The investigational medical devices (IMDs) of the planned clinical evaluation, Leukomed® T skin sensitive and Leukomed® T plus skin sensitive have been developed for treatment of acute wounds on patients with fragile or sensitive skin to provide a reliable but skin-friendly fixation and wound care option.

The primary purpose of this clinical study is the evaluation of clinical performance to stay in place up to seven days and the safety of both dressings. Further, data on wearing comfort, product handling, pain during removal and quality of life are considered as secondary outcomes. The products will be used as part of routine wound care within the scope of their intended purpose without any additional invasive or burdensome examination.

ELIGIBILITY:
Inclusion Criteria:

* Men, women or diverse
* ≥ 65 years of age
* Patient is mentally and physically able to participate in this study
* Signed informed consent to participate in this study
* Fragile skin condition
* Acute wound (surgical wound or laceration), indicated for treatment with the investigational products for a time period of 7 days

Exclusion Criteria:

* Infection of the target wound
* Alcohol or drug addiction
* Known sensitivity or allergy to any component of the study product
* Patients who participate in any other clinical study investigating drugs or medical devices

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Subjects 65 years and older suffering from skin changes causing fragile skin. Extrinsic factors and intrinsic factors leading to skin damages or pathological changes: extremes of ager (>80 years), race/ethnicity, underlaying medical conditions, dermatological conditions, malnutrition, dehydration, drying of the skin, prolonged exposure to moisture, certain medication, current radiotherapy, photedamage, previous removal of tapes/dressings/devices, repeated taping. Subject presenting on of the criteria above can be included.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Adhered dressing area after wear | 7 days after dressing application
  Percentage of adhered dressing area 7 days after application

SECONDARY OUTCOMES:
Skin damage | 7 days after dressing application
  skin damage after dressing removal
Skin reddening | 7 days after dressing application
  Reddening of the skin 30 min after dressing removal
Skin reactions | after 7 days
  Further skin reactions after dressing removal
Pain assessment | 7 days after dressing application
  Pain at dressing removal
Product Evaluation by patient | 7 days after dressing application
  Judge wearing comfort
Product Evaluation by Health Care Professional | at application day (day 0)
  Assessment of handling, application and and re-application
Infection | 7 days after dressing application
  Assess signs of wound infection

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Practice Degenhardt, Bremen
  - Klinikum Dortmund, Dortmund
  - orthoGroup, Hamburg

IPD SHARING:
Plan to Share IPD: No
data will not be shared